CLINICAL TRIAL: NCT03200119
Title: A Study of the Management of the Patient's Disease Based on the Life Log Data of Patients With Lifestyle-related Diseases Through a Wearable Device
Brief Title: MyHealthKeeper: Clinical Trial Study Based on Personal Health Record Healthcare Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Se Young Jung, Clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1504/296-302
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application user group (Experimental): In the active group, participants were educated to modify their lifestyle to lose weight by using a smart phone-based lifestyle app which was designed to collect daily activity and dietary information. The app was composed of two main modules: a diet module, and a physical activity module.
  Interventions: Behavioral: Daily health-related lifestyle modification prescription
- Control group (No Intervention): Conventional lifestyle modification

INTERVENTIONS:
Behavioral: Daily health-related lifestyle modification prescription — Daily health-related lifestyle modification prescription
  Arms: Mobile application user group

SUMMARY:
In order to study the effectiveness of personalized healthcare intervention for lifestyle-related diseases, investigators designed this study using mobile application and clinical feedback from clinicians

ELIGIBILITY:
Inclusion Criteria:

* Study participants must agree to support by him/herself at enroll time
* Patients without severe cardiopulmonary disease, cancer, or other acute diseases
* Patients must be over BMI > 23 kg/m2

Exclusion Criteria:

* Patient who did not agree with this study
* Patients with severe cardiopulmonary disease, cancer, or other acute diseases
* Patients who were pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Body weight change | baseline and after 4weeks of lifestyle intervention
  weight measurement and calculate BMI(body mass index)

SECONDARY OUTCOMES:
Blood test result change | baseline and after 4weeks of lifestyle intervention
  Blood test and its several results value measurement
Mobile-app usage change | baseline and after 4weeks of lifestyle intervention
  Usage log of mobile application

CONTACTS AND LOCATIONS:
Overall Officials: Se young Jung, MD, MPH, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No
patient personal information is confidential according to the hospital's data protection policy

REFERENCES:
- [Derived] Ryu B, Kim N, Heo E, Yoo S, Lee K, Hwang H, Kim JW, Kim Y, Lee J, Jung SY. Impact of an Electronic Health Record-Integrated Personal Health Record on Patient Participation in Health Care: Development and Randomized Controlled Trial of MyHealthKeeper. J Med Internet Res. 2017 Dec 7;19(12):e401. doi: 10.2196/jmir.8867. PMID 29217503